CLINICAL TRIAL: NCT03515954
Title: Anterior Segment Optical Coherence Tomography (AS-OCT) Guided Treatment of Diffuse Conjunctival Squamous Cell Carcinoma (CSCC) With Excision, Amniotic Membrane Graft Using Fibrin Glue and Topical Mitomycin C (MMC)
Brief Title: AS-OCT Guided Treatment of Diffuse CSCC
Status: Completed | Type: Observational
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Tarek Roshdy mohamed Mahgoub ELhamaky, lecturer of ophthalmology, Benha University
Other Study IDs: benha19992
Record Dates: First submitted 2018-04-24; First posted 2018-05-04 (Actual); Last update posted 2019-01-02 (Actual); Status verified 2018-12

CONDITIONS: Conjunctival Neoplasms
Keywords: conjunctiva; squamous neoplasia; amniotic
MeSH Terms: conditions — Conjunctival Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Treatment of diffuse ocular surface squamous neoplasia — Excision of the conjunctival tumour was done.Amniotic membrane was secured into conjunctival defects. Postoperative topical MMC 0.04% was given. Response to treatment was monitored clinically and by AS-OCT.

SUMMARY:
A prospective study was performed on 8 eyes of 8 patients who underwent amniotic membrane graft after diffuse conjunctival squamous cell neoplasia excision followed by topical mitomycin C 0.04% eye drop between March 2014 and January 2018.

DETAILED DESCRIPTION:
Surgical excision of the conjunctival tumour . A superficial corneal scraping was performed for corneal lesion then double freeze-thaw cryotherapy was applied to limbal edge and conjunctival margins.The amniotic membrane graft was secure and attached to the sclera and conjunctiva using ﬁbrin glue.Topical mitomycin C 0.04%eye drop was prescribed 4 times daily per treatment cycle (1 cycle=1 week on 1 week off).

ELIGIBILITY:
Inclusion Criteria:

* diffuse Ocular Surface Squamous Neoplasia

Exclusion Criteria:

* localized OSSN (less than ﬁve clock hours in limbal extent)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study included 8 eyes of 8 patients. The mean age of all patients was 51.9 ± 9.9 years. There were 7 males (87.5%) and 1 female (12.5%).
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
The recurrence rate of lesion | 2 years
  Any recurrence which is detected clinically or/and by AS-OCT